CLINICAL TRIAL: NCT07284160
Title: A Study on the Effectiveness of Rest Shame Interventions Based on Cognitive Behavioural Therapy in Reducing Social Media Addiction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: KY-2025-286
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Rest is Shameful

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured intervention based on cognitive behavioural therapy (CBT) (Experimental): Structured intervention based on cognitive behavioural therapy (CBT)
  Interventions: Other: Structured intervention based on cognitive behavioural therapy (CBT)
- Control group (No Intervention)

INTERVENTIONS:
Other: Structured intervention based on cognitive behavioural therapy (CBT) — Structured intervention based on cognitive behavioural therapy (CBT)
  Arms: Structured intervention based on cognitive behavioural therapy (CBT)

SUMMARY:
This study will employ a randomised controlled trial design to systematically intervene in university students' rest shaming through a structured intervention programme grounded in cognitive behavioural therapy (CBT), thereby examining its efficacy in reducing social media addiction. Through this research, we aim to evaluate the effectiveness of CBT interventions in alleviating rest shaming and demonstrate that operationalising rest shaming influences social media addiction.

ELIGIBILITY:
Inclusion Criteria:

* University students aged 18-25 who are capable of understanding and completing research-related tasks, and who have confirmed the presence of rest shaming experiences via the Rest Shaming Scale.

Exclusion Criteria:

* Individuals with a history of severe mental illness (such as clinically diagnosed depression, anxiety disorders, etc.), cognitive impairment, or an inability to cooperate in completing the research process.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
rest intolerance scale | From enrollment to the end of treatment at 1 week
Social media addiction | From enrollment to the end of treatment at 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Yiwu, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No